CLINICAL TRIAL: NCT02827565
Title: Prospective Study of Technical Optimization of the Detection of KRAS Mutations, BRAF and NRAS by Next Generation Sequencing on Tumor DNA Circulating in Metastatic Colorectal Cancer.
Brief Title: Technical Optimization of Detection of KRAS, BRAF and NRAS Mutations on Tumor DNA Circulating in Metastatic Colorectal Cancer
Acronym: CircuLOR-1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut de Cancérologie de Lorraine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2015-A00922-47
Record Dates: First submitted 2016-07-06; First posted 2016-07-11 (Estimated); Last update posted 2018-08-08 (Actual); Status verified 2018-08

CONDITIONS: Metastatic Colorectal Cancer
Keywords: colorectal cancer; Kras mutation; Nras mutation; Braf mutation
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CircuLOR-1 (Experimental): KRAS (exons 2, 3 et 4), NRAS (exons 2, 3 et 4) and BRAF (exon 15) mutations
  Interventions: Other: KRAS, NRAS et BRAF mutation analysis from circulating plasma DNA

INTERVENTIONS:
Other: KRAS, NRAS et BRAF mutation analysis from circulating plasma DNA — 10 ml blood sample
  Other Names: NGS

SUMMARY:
The objective of this study is to optimize the search by next-generation sequencing (NGS) mutations in the KRAS, BRAF and NRAS on circulating tumor DNA and compare the genetic profiles obtained with those from tumors embedded in paraffin

ELIGIBILITY:
Inclusion Criteria:

* Patients with metastatic or locally advanced colorectal carcinoma with a KRAS, BRAF or NRAS mutation
* Age ≥ 18 years
* Patient information and written informed consent form signed
* Patient must be affiliated to a social security system

Exclusion Criteria:

* Patients whose health-cons indicates a blood sample 10mL
* Age < 18 years
* Pregnant or breast feeding females
* Persons deprived of liberty or under supervision

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-02-03 (Actual); Primary Completion 2017-01-05 (Actual); Study Completion 2017-01-19 (Actual)

PRIMARY OUTCOMES:
Technical Optimization of KRAS, BRAF and NRAS mutations detection | 1 day
  Optimize the detection of mutations of KRAS (exons 2, 3 et 4), NRAS (exons 2, 3 et 4) and BRAf (exon 15) genes, using the next-generation sequencing technology from circulating tumor DNA in patients with metastatic colorectal cancer.

SECONDARY OUTCOMES:
KRAS, NRAS et BRAF mutational status | 1 day
  Compare the results of KRAS NRAS and BRAF genes genotyping obtained from circulating tumor DNA to that achieved by the current gold standard (paraffin-embedded).

CONTACTS AND LOCATIONS:
Overall Officials: GAVOILLE CELINE, MD, Principal Investigator — Institut de Cancérologie de Lorraine; HARLE ALEXANDRE, Study Chair — Institut de Cancérologie de Lorraine
Locations (1):
- Institut de Cancerologie de Lorraine, Vandœuvre-lès-Nancy, France

IPD SHARING:
Plan to Share IPD: No